CLINICAL TRIAL: NCT01434355
Title: Molecular Epidemiology of Pediatric Germ Cell Tumors
Brief Title: DNA Analysis in Samples From Younger Patients With Germ Cell Tumors and Their Parents or Siblings
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AEPI10N1; NCI-2011-03464 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000711070; COG-AEPI10N1; AEPI10N1 (Other: Childrens Oncology Group); AEPI10N1 (Other: CTEP)
Record Dates: First submitted 2011-09-13; First posted 2011-09-14 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2017-10

CONDITIONS: Childhood Malignant Ovarian Germ Cell Tumor; Childhood Malignant Testicular Germ Cell Tumor; Ovarian Choriocarcinoma; Ovarian Embryonal Carcinoma; Ovarian Mixed Germ Cell Tumor; Ovarian Teratoma; Ovarian Yolk Sac Tumor; Testicular Choriocarcinoma; Testicular Embryonal Carcinoma; Testicular Seminoma; Testicular Teratoma; Testicular Yolk Sac Tumor
MeSH Terms: conditions — Ovarian Germ Cell Cancer; Testicular Neoplasms; Teratoma, Ovarian; Seminoma; Teratoma, Testicular; Endodermal Sinus Tumor

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva and tissue

GROUPS / COHORTS (1):
- Correlative studies: Patients and parents or siblings undergo saliva sample collection. DNA extracted from saliva samples and from patients' archived tumor tissue samples is genotyped and analyzed by methylation arrays, including methylation-specific PCR (pyrosequencing) assays. Genetic variation between pediatric germ cell tumors and parent or sibling is also analyzed. Patients' and family members' health history, demographics, and environmental exposures are collected by questionnaires or telephone interviews. Medical history, such as chronic conditions, prescribed medications and congenital abnormalities, including cryptorchidism, is also collected. Birth characteristics of the child, including birth weight and gestational age, are also captured.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This research trial studies deoxyribonucleic acid (DNA) samples from younger patients with germ cell tumor and their parents or siblings. Studying samples of tumor tissue and saliva from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To evaluate associations between genetic variation and pediatric germ cell tumor (GCT) using a case-parent triad design to identify variants in four genes, KITLG, SPRY4, BAK1, and DMRT1, associated with pediatric GCT.

II. To evaluate associations between genetic variation and pediatric GCT using a case-parent triad design to include targeted genotyping of single nucleotide polymorphisms (SNPs) in selected key pathways essential for normal in utero germ cell development, specifically genes involved in survival of germ cells during migration, apoptosis, and cell cycle control.

III. To explore inter- and intratumoral heterogeneity in DNA methylation by tumor histology.

OUTLINE: This is a multicenter study.

Patients and parents or siblings undergo saliva sample collection. DNA extracted from saliva samples and from patients' archived tumor tissue samples is genotyped and analyzed by methylation arrays, including methylation-specific polymerasechain reaction (PCR) (pyrosequencing) assays. Genetic variation between pediatric germ cell tumors and parent or sibling is also analyzed. Patients' and family members' health history, demographics, and environmental exposures are collected by questionnaires or telephone interviews. Medical history, such as chronic conditions, prescribed medications and congenital abnormalities, including cryptorchidism, is also collected. Birth characteristics of the child, including birth weight and gestational age, are also captured.

ELIGIBILITY:
Inclusion Criteria:

* The patient is enrolled on COG-ACCRN07
* The patient has a primary diagnosis of germ cell tumor (GCT) including germinoma (ICCC 9060-9065) teratoma (9080-9084), embryonal carcinoma (9070-9072), yolk sac tumor (9071),choriocarcinoma (9100, 9103, 9104), and mixed GCT (9085, 9101, 9102, 9105) in all sites including the brain and central nervous system and registered with Children's Oncology Group (COG) by a North American member institution
* The patient must be diagnosed with a germ cell tumor between July 1, 2008 and December 31, 2015
* The patient must be < 20 years of age at the time of diagnosis
* The patient must have at least one biological parent alive and willing to participate

  * In the event that one case parent cannot contribute DNA, a case sibling, defined as the biological brother or sister of the study subject, may donate instead
* All questionnaire respondents must understand English or Spanish
* Concomitant treatment on a therapeutic trial is not required

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Sampling Method: Non-Probability Sample
Enrollment: 932 (Estimated)
Dates: Start 2011-11-01 (Actual); Primary Completion 2016-08-04 (Actual); Study Completion 2016-08-04 (Actual)

PRIMARY OUTCOMES:
Pediatric GCT associated with genetic susceptibility | Up to 5 years
  Will be modeled using a Poisson regression. A likelihood ratio test determines the statistical significance.

SECONDARY OUTCOMES:
List of genes that distinguish between the three most common histologic subtypes of pediatric GCT: yolk sac tumor, teratoma, and germinoma | Up to 5 years
  A permutation based Chi-Square test for categorical covariates or a permutation based Kruskal-Wallis test (continuous risk factors) will be used.
Validation of array results by pyrosequencing | Up to 5 years
  A standard case-only approach evaluating differences in methylation by histology, age and gender will be done using chi-square and ANOVA.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Poynter, Principal Investigator — Children's Oncology Group
Locations (1):
- Childrens Oncology Group, Philadelphia, Pennsylvania, United States